CLINICAL TRIAL: NCT06809023
Title: Evaluation of Sex Differences in Glucose Metabolism in Response to Sleep Curtailment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Charles A. Czeisler, PhD, MD, Professor of Sleep Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2025-P-000064
Record Dates: First submitted 2025-01-24; First posted 2025-02-05 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Sleep Deprivation; Sex Differences; Glucose Tolerance
Keywords: glucose metabolism; sleep deprivation; sex differences; GLP-1
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: This study uses a within-subjects randomized crossover design to compare the effects of sleep restriction to a control condition where participants are not sleep restricted.
Who Masked: Participant
Masking Description: The order in which participants complete the study arms is randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep restriction (Experimental): Participants undergo sleep restriction to 4 hours/night
  Interventions: Behavioral: Sleep restriction
- Control condition (No Intervention): Participants undergo the control condition (no sleep restriction)

INTERVENTIONS:
Behavioral: Sleep restriction — Participants will be asked to sleep 4h/night
  Arms: Sleep restriction

SUMMARY:
The goal of this study is to learn whether insufficient sleep affects glucose metabolism differently in healthy men and women.

DETAILED DESCRIPTION:
Two-thirds of Americans report regularly obtaining an insufficient amount of sleep. Chronic sleep deficiency is associated with negative health consequences such as obesity, cardiovascular disease, diabetes, and metabolic syndrome. Laboratory studies have shown that sleep restriction reduces glucose tolerance in otherwise healthy adults, and it is now well established that sleep restriction decreases insulin sensitivity. However, there is a significant gap in the literature regarding how sex differences may drive disparate metabolic outcomes in men and women in response to sleep loss.

Epidemiological studies strongly suggest that women and men may respond differently to the physiological challenges associated with sleep restriction and circadian disruption. Trouble sleeping is more prevalent in women compared to men, and sleep disturbances appear to be associated with higher risk of obesity, hypertension, and elevated HbA1c in women compared to men. Although multiple causative mechanisms have been explored, most laboratory studies investigating the mechanisms by which sleep disturbances impair metabolism have been conducted solely in men or have not been powered for sex differences.

One potential mechanism underlying sex differences in glucose regulation after sleep loss is the glucagon-like peptide-1 (GLP-1) pathway. GLP-1 reduces blood glucose by stimulating insulin secretion and inhibiting glucagon secretion in response to food intake and is the target of promising new treatments for insulin resistance and obesity such as Ozempic and Wegovy. Interestingly, women exhibit a greater response to treatment with these GLP-1 receptor agonist drugs; additionally, one laboratory study found decreased GLP-1 levels in women but not in men after 4 days of sleep curtailment.

This study will use a randomized crossover design in young men and premenopausal women to test the hypotheses that sleep loss impairs glucose tolerance more in women than in men, and that this difference is partially mediated by sex-dependent responses in GLP-1 after sleep curtailment.

Currently, there are no sex-specific recommendations for management of diabetes or sleep loss, despite evidence that women may bear a greater disease burden than men. Understanding sex differences in glucose metabolism in response to sleep curtailment is critical for making more effective and individualized treatment recommendations to mitigate the adverse metabolic effects of sleep restriction in women and men.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults with conventional sleep-wake timing
* Non-smokers
* Completion of medical, psychological, and sleep screening tests
* Able to spend 5 consecutive days/nights in the laboratory on two separate occasions (total of 10 days/nights in the laboratory)
* Women must have a recent history of regular menstrual cycles

Exclusion Criteria:

* History of neurological or psychiatric disorder
* History of sleep disorder or regular use of sleep-promoting medication
* Current prescription, herbal, or over-the-counter medication use including hormonal birth control
* Traveling across 2 or more time zones within past 3 months
* Donating blood within past 8 weeks
* Worked night or rotating shift work within past year
* Hearing impairment, visual impairment
* History of eye trauma or surgery
* Drug or alcohol dependency

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — At this time, we are recruiting cisgender men and women
Enrollment: 32 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Difference between men and women in postprandial glucose response after Sleep Restriction | Study Day 4 (Arm 1) vs. Study Day 4 (Arm 2)
  Test the hypothesis that three nights of sleep curtailment increases postprandial glucose levels to a greater extent in women compared to men. Postprandial glucose will be assessed in response to a standard meal after Control and Sleep Restriction. The change in postprandial glucose from Control to Sleep Restriction will be compared between men and women.
Difference between men and women in postprandial GLP-1 response after Sleep Restriction | Study Day 4 (Arm 1) vs. Study Day 4 (Arm 2)
  Test the hypothesis that three nights of sleep curtailment decreases postprandial GLP-1 levels to a greater extent in women compared to men. Postprandial GLP-1 levels will be assessed in response to a standard meal after Control and Sleep Restriction. The change in postprandial GLP-1 from Control to Sleep Restriction will be compared between men and women.

SECONDARY OUTCOMES:
Difference between men and women in fasting glucose after Sleep Restriction | Study Day 5 (Arm 1) vs. Study Day 5 (Arm 2)
  Test the hypothesis that three nights of sleep curtailment increases fasting glucose levels to a greater extent in women compared to men. Fasting glucose will be assessed overnight during the habitual sleep period after Control and Sleep Restriction. The change in fasting glucose from Control to Sleep Restriction will be compared between men and women.
Difference between men and women in fasting GLP-1 after Sleep Restriction | Study Day 5 (Arm 1) vs. Study Day 5 (Arm 2)
  Test the hypothesis that three nights of sleep curtailment decreases fasting GLP-1 levels to a greater extent in women compared to men. Fasting GLP-1 levels will be assessed overnight during the habitual sleep period after Control and Sleep Restriction. The change in fasting GLP-1 from Control to Sleep Restriction will be compared between men and women.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No